CLINICAL TRIAL: NCT05115786
Title: Cohort Study to Evaluate the Relapse Risk Test in Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HBI Solutions Inc. (Industry)
Collaborators: mProbe Inc. (Industry)
Responsible Party: Principal Investigator, Junjie Peng, Professor, Shanghai Cancer Hospital, China
Other Study IDs: CRC_Relapse_001
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — FFPE
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort A: FFPE specimen collection. FFPE tumor tissue samples must be collected after surgical resection and before starting chemotherapy or other treatment.
- Cohort B: FFPE specimen collection. FFPE tumor tissue samples must be collected after surgical resection and before starting chemotherapy or other treatment.
- Cohort C: FFPE specimen collection. FFPE tumor tissue samples must be collected after surgical resection and before starting chemotherapy or other treatment.
- Cohort D: FFPE specimen collection. FFPE tumor tissue samples must be collected after surgical resection and before starting chemotherapy or other treatment.

SUMMARY:
A Retrospective Cohort Study to Evaluate a Multigene assay to assess the recurrence risk of colorectal cancer.

DETAILED DESCRIPTION:
Colon cancer is the fourth most prevalent cancer for both men and women and also the third most common cause of cancer-related deaths worldwide. The primary consideration in deciding whether the moderate benefits from adjuvant chemotherapy for colon cancer (a 20% to 25%proportional reduction in the risk of recurrence and death) will be worth-while is the likelihood of disease recurrence, with larger absolute benefits for higher-risk patients. Nevertheless, the recurrence of cancer and decisions about its treatment still rely largely on classic histopathological and immuno histochemical techniques.

The purpose of this study is to validate a previously developed multigene assay for a more quantitative approach to predict the recurrence risk and rational individualization of treatment are needed. A retrospective cohort of stage II and stage III patients with average 5 years follow up after resection surgery will be selected. Formalin fixed paraffin-embedded (FFPE) tumor tissue collected during patients' resection surgery with either recurrence or non-recurrence follow-up will be used validate the test. This multigene assay result will provide a precise estimate of the risk of recurrence and chemotherapy benefit for colorectal patients to help guide the most appropriate treatment decision.

Three types of patients in this study:

Cohort A

People ages 20 year or older who were diagnosed with anatomic stage II, T3, MMR-P colorectal cancer and had recurrence of tumor within 5 years follow-up. FFPE tumor tissue samples must be collected after surgical resection and before starting chemotherapy or other treatment.

Cohort B

People ages 20 year or older who were diagnosed with anatomic stage II, T3, MMR-P colorectal cancer and had no-recurrence of tumor within 5 years follow-up. FFPE tumor tissue samples must be collected after surgical resection and before starting chemotherapy or other treatment.

Cohort C

People ages 20 year or older who were diagnosed with stage III A/B colorectal cancer and had recurrence of tumor within 5 years follow-up. FFPE tumor tissue samples must be collected after surgical resection and before starting chemotherapy or other treatment.

Cohort D

People ages 20 year or older who were diagnosed with stage III A/B colorectal cancer and had no-recurrence of tumor within 5 years follow-up. FFPE tumor tissue samples must be collected after surgical resection and before starting chemotherapy or other treatment.

ELIGIBILITY:
Cohort A

Inclusion Criteria:

* Subjects must be 20 years of age or older.
* Subjects was diagnosed with anatomic stage II, T3, MMR-P colorectal cancer
* Subjects had recurrence date information within 5 years follow-up after initial tumor resection surgery
* Subject is able and willing to provide FFPE sample per protocol
* Subject is able to comprehend and willing to sign and date the written informed consent document(s) and any applicable medical record release documents for the study

Exclusion Criteria:

* No tumor block available from initial diagnosis before any chemotherapy treatment
* Presence of synchronous tumors
* No tumor or very little tumor (<5% tumor present) in block as assessed designated pathologist.
* Tumor types other than adenocarcinoma NOS (not otherwise specified) and mucinous carcinoma as assessed by examination of the H&E slide by designated pathologist.
* Insufficient RNA (<5 ng/μL or 300 ng) for RT-PCR analysis.
* Failure of assay to meet pre-specified quality control (QC) specifications.

Cohort B

Inclusion Criteria:

* Subjects must be 20 years of age or older.
* Subjects was diagnosed with anatomic stage II, T3, MMR-P colorectal cancer
* Subjects had 5 years follow-up information after initial tumor resection surgery
* Subject is able and willing to provide FFPE sample per protocol
* Subject is able to comprehend and willing to sign and date the written informed consent document(s) and any applicable medical record release documents for the study

Exclusion Criteria:

* No tumor block available from initial diagnosis before any chemotherapy treatment
* Presence of synchronous tumors
* No tumor or very little tumor (<5% tumor present) in block as assessed designated pathologist.
* Tumor types other than adenocarcinoma NOS (not otherwise specified) and mucinous carcinoma as assessed by examination of the H&E slide by designated pathologist.
* Insufficient RNA (<5 ng/μL or 300 ng) for RT-PCR analysis.
* Failure of assay to meet pre-specified quality control (QC) specifications.

Cohort C

Inclusion Criteria:

* Subjects must be 20 years of age or older.
* Subjects was diagnosed with anatomic stage III A/B colorectal cancer
* Subjects had recurrence date information within 5 years follow-up after initial tumor resection surgery
* Subject is able and willing to provide FFPE sample per protocol
* Subject is able to comprehend and willing to sign and date the written informed consent document(s) and any applicable medical record release documents for the study

Exclusion Criteria:

* No tumor block available from initial diagnosis before any chemotherapy treatment
* Presence of synchronous tumors
* No tumor or very little tumor (<5% tumor present) in block as assessed designated pathologist.
* Tumor types other than adenocarcinoma NOS (not otherwise specified) and mucinous carcinoma as assessed by examination of the H&E slide by designated pathologist.
* Insufficient RNA (<5 ng/μL or 300 ng) for RT-PCR analysis.
* Failure of assay to meet pre-specified quality control (QC) specifications.

Cohort D

Inclusion Criteria:

* Subjects must be 20 years of age or older.
* Subjects was diagnosed with anatomic stage III A/B colorectal cancer
* Subjects had 5 years follow-up information after initial tumor resection surgery
* Subject is able and willing to provide FFPE sample per protocol
* Subject is able to comprehend and willing to sign and date the written informed consent document(s) and any applicable medical record release documents for the study

Exclusion Criteria:

* No tumor block available from initial diagnosis before any chemotherapy treatment
* Presence of synchronous tumors
* No tumor or very little tumor (<5% tumor present) in block as assessed designated pathologist.
* Tumor types other than adenocarcinoma NOS (not otherwise specified) and mucinous carcinoma as assessed by examination of the H&E slide by designated pathologist.
* Insufficient RNA (<5 ng/μL or 300 ng) for RT-PCR analysis.
* Failure of assay to meet pre-specified quality control (QC) specifications.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is an exploratory study utilizing archived tumor specimens and demographic and pathologic characteristics derived from the patient's medical charts. As such, all eligible patients must have a stored tumor specimen which can be accessed for analysis.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of colorectal cancer | 5 years
  Recurrence of anatomic stage II, MMR-P and stage III A/B colorectal patients

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Peng, M.D, Principal Investigator — Shanghai Cancer Hospital, China

IPD SHARING:
Plan to Share IPD: Undecided